CLINICAL TRIAL: NCT04227171
Title: A Multicenter, Prospective Cohort Observational Study to Develop Dosing Chart Based on Patient Specific Characteristics and Ovarian Response When Follitrope™ PFS is Administered Subcutaneously to Infertility Women Patients
Brief Title: Observational Study to Develop Dosing Chart
Status: Completed | Type: Observational
Sponsor: LG Chem (Industry)
Responsible Party: Sponsor
Other Study IDs: LG-FSOS002
Record Dates: First submitted 2020-01-05; First posted 2020-01-13 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Infertile Women Undergoing IVF or ICSI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Weeks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- FSH only: GnRH agonist protocol & GnRH antagonist protocol

SUMMARY:
To confirm the predictors based on patient specific characteristics and ovarian response and develop dosing chart when Follitrope™ PFS is administered to infertility women patients.

ELIGIBILITY:
Inclusion Criteria:

* Female aged of 19 to 39 years
* Mean menstrual cycle in 25 to 35 days
* Patients to whom Follitrope PFS will be administered in those scheduled to undergo the IVF-ET according to the GnRH agonist or antagonist protocol
* In the past continuous IVF cycle failure less than 2 times

Exclusion Criteria:

* Patients having a history of ovarian, breast, uterus, hyperthalamus, or pituitary tumor
* Abnormal uterine bleeding of undetermined origin
* Prior hypersensitivity to a component of recombinant FSH
* Ovarian cyst or enlargement of undetermined origin
* Clinically significant endocrine abnormalities
* Patients having polycystic ovary syndrome (PCOS) history
* Poor Ovarian responder (Bologna criteria)
* Patients who received Clomiphene citrate, Letrozole (Pemara), or Gonadotropin within 30 days prior to enrollment in this study

Ages: 19 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Infertile women undergoing In vitro fertilization(IVF) or Intracytoplasmic sperm injection (ICSI) for controlled ovarian stimulation
Sampling Method: Probability Sample
Enrollment: 534 (Actual)
Dates: Start 2018-08-03 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
No. of oocytes retrieved No. of oocytes retrieved Number of oocyte retrieved | after OPU, normally 2 weeks
  Number of oocyte identified by ovum pick up (OPU) after overovulation

SECONDARY OUTCOMES:
Oocyte maturity quality | after OPU, normally 2 weeks
  Metaphase II oocytes (%, ICSI only)
Total dose (IU) of Follitrope™ PFS administered | 2 weeks
Total duration (days) of Follitrope™ PFS administered | 2 weeks
E2 concentration on hCG day | normally 10 days
P4 concentration on hCG day | normally 10 days
Fertilization rate | 1~2 days after OPU
Number of embryo transferred | 3~5 days after OPU
Implantation rate | 24 days after OPU
Biochemical pregnancy rate | 10 days after OPU
clinical pregnancy rate | 24 days after OPU
pregnancy rate | up to 10 weeks after OPU

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul Maria Fertility Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No